CLINICAL TRIAL: NCT05830123
Title: ARTEMIS-002: A Phase 2, Multicenter, Open-label Study of Intravenous Administration of HS-20093 in Patients With Relapsed or Refractory Osteosarcoma and Other Sarcomas
Brief Title: ARTEMIS-002: HS-20093 in Patients With Relapsed or Refractory Osteosarcoma and Other Sarcomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20093-201
Record Dates: First submitted 2023-04-03; First posted 2023-04-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Osteosarcoma; Sarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort 1 at HS-20093 8mg/kg (Phase 2a) (Experimental): Participants in cohort 1 will be randomized to receive HS-20093 at 8 mg/kg.
  Interventions: Drug: HS-20093
- cohort 1 at HS-20093 12mg/kg (Phase 2a) (Experimental): Participants in cohort 1 will be randomized to receive HS-20093 at 12 mg/kg.
  Interventions: Drug: HS-20093
- cohort 2 at HS-20093 12mg/kg (Phase 2a) (Experimental): Participants in cohort 2 will receive HS-20093 at 12 mg/kg.
  Interventions: Drug: HS-20093
- HS-20093(Phase 2b) (Experimental): Participants will receive HS-20093 at the recommended dose from Phase 2a.
  Interventions: Drug: HS-20093

INTERVENTIONS:
Drug: HS-20093 — IV administration of HS-20093 Q3W; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.

SUMMARY:
HS-20093 is a fully humanized IgG1 antibody-drug conjugate (ADC) which specifically binds to B7-H3, a target wildly expressed on solid tumor cells.

This is a phase 2, open-label, multi-center study to evaluate the efficacy, safety, pharmacokinetics (PK) and immunogenicity of HS-20093 as a monotherapy in patients with relapsed or refractory osteosarcoma and other sarcomas.

DETAILED DESCRIPTION:
This is a phase 2, open-label, multi-center study consisting of two parts: Phase 2a and 2b.

Phase 2a: The study will be conducted in the following two cohorts: Cohort 1: Patients with advanced osteosarcoma upon disease progression after standard treatment. Cohort 2: Patients with other unresectable bone and soft tissue sarcomas, if they have progressed on or intolerant to available standard therapies, or no standard or available curative therapy exists. Subjects will be randomly assigned in a 1:1 ratio to 8.0 mg/kg and 12.0 mg/kg of HS-20093 in cohort 1 and will receive 12.0 mg/kg in cohort 2.

Phase 2b: The study will be conducted in patients with advanced osteosarcoma upon disease progression after standard treatment. Subjects will receive HS-20093 at the recommended dose from Phase 2a.

All patients will be carefully followed for adverse events during the study treatment and for 90 days after the last dose of HS-20093. Subjects will be permitted to continue therapy with assessments for progression if the product is well tolerated and sustained clinical benefit exists.

ELIGIBILITY:
Inclusion Criteria:

1. At least age of 18 years at screening;
2. Patients with histologically confirmed relapsed or refractory osteosarcoma or other sarcomas who have progressed upon first-line systemic treatment.
3. At least one measurable lesion according to RECIST 1.1.
4. Agree to provide fresh or archival tumor tissue and peripheral blood samples.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1
6. Life expectancy >= 12 weeks
7. Men or women should be using adequate contraceptive measures throughout the study;
8. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential
9. Signed and dated Informed Consent Form

Exclusion Criteria:

1. Treatment with any of the following:

   1. Previous or current treatment with B7-H3 targeted therapy
   2. Any cytotoxic chemotherapy, investigational agents and anticancer drugs within 14 days prior to the first scheduled dose of HS-20093
   3. Prior treatment with a monoclonal antibody within 28 days prior to the first scheduled dose of HS-20093
   4. Radiotherapy with a limited field of radiation for palliation within 2 weeks, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks prior to the first scheduled dose of HS-20093
   5. Pleural or peritoneal effusion requiring clinical intervention. Pericardial effusion.
   6. Major surgery within 4 weeks of the first dose of HS-20093.
   7. Spinal cord compression or brain metastases.
   8. Treatment with drugs that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug; or requiring treatment with these drugs during the study.
   9. Currently receiving drugs known to prolong QT interval or may cause torsade de pointe; or requiring treatment with these drugs during the study.
2. Any unresolved toxicities from prior therapy greater than Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0 with the exception of alopecia or neurotoxicity.
3. History of other primary malignancies.
4. Inadequate bone marrow reserve or organ dysfunction
5. Evidence of cardiovascular risk.
6. Severe, uncontrolled or active cardiovascular diseases.
7. Diabetes ketoacidosis or hyperglycemia hypertonic occurring within 6 months before the first dose of the study drug, or the glycosylated hemoglobin value ≥ 7.5% in the screening period.
8. Severe or poorly controlled hypertension.
9. Bleeding symptoms with apparent clinical significance or obvious bleeding tendency within 1 months prior to the first dose of HS-20093
10. Serious arteriovenous thrombosis events occurred within 3 months before the first dose.
11. Severe infections occurred within 4 weeks before the first dose.
12. Patients who have received continuous steroid treatment for more than 30 days within 30 days before the first dose, or need long-term (≥ 30 days) steroid treatment, or who have other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation
13. The presence of active infectious diseases has been known before the first dose such as hepatitis B, hepatitis C, tuberculosis, syphilis, or human immunodeficiency virus HIV infection, etc.
14. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh Grade B or more severe cirrhosis.
15. Other moderate or severe lung diseases that may interfere with the detection or treatment of drug-related pulmonary toxicity or may seriously affect respiratory function.
16. Previous history of serious neurological or mental disorders, including epilepsy, dementia or severe depression and any other status that may interfere in assessment.
17. Women who are breastfeeding or pregnant or planned to be pregnant during the study period.
18. Vaccination or hypersensitivity of any level within 4 weeks prior to the first dose of HS-20093
19. History of severe hypersensitivity reaction, severe infusion reaction or allergy to recombinant human or mouse derived proteins.
20. Hypersensitivity to any ingredient of HS-20093.
21. Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator
22. Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) determined by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | From the first dose up to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigators based on RECIST version 1.1[Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From the first dose through 90 days post end of treatment.
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a clinical study participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.
Observed maximum plasma concentration (Cmax) of HS-20093 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Cmax will be obtained following administration of the first dose of HS-20093 during the first cycle.
Time to reach maximum plasma concentration (Tmax) of HS-20093 following the first dose | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Tmax will be obtained following administration of the first dose of HS-20093 during the first cycle.
Terminal half-life (T1/2) of HS-20093 following the first dose | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-20093 | From pre-dose to 14 days after the first dose on Cycle 1 (each cycle is 21 days)
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Percentage of participants with antibodies to HS-20093 in serum | From pre-dose to 90 days post end of treatment
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points.
ORR determined by Independent review committee (IRC) according to RECIST 1.1 | From the first dose up to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by IRC based on RECIST version 1.1[Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Duration of response (DoR) determined by investigators and IRC according to RECIST 1.1 | From the first dose up to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  DoR was defined as the period from the first occurrence of CR or PR to progressive disease (PD) or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Disease control rate (DCR) determined by investigators and IRC according to RECIST 1.1. | From the first dose up to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks); SD shall be assessed at least 5 weeks after the first dose].
Progression-free survival (PFS) determined by investigators and IRC according to RECIST 1.1 | From the first dose or random assignment up to disease progression or withdrawal from study, whichever came first, assessed up to 24 months.
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). PFS was defined as the time from first dose or random assignment (if any) to PD or death from any cause.
4-month PFS rate determined by investigators and IRC according to RECIST 1.1 | 4 months.
  4-month PFS rate is defined as the percentage of patients whose disease is progression free at 4 months from the start of treatment.
Overall survival (OS) | From the first dose or random assignment up to death or withdrawal from study, whichever came first, assessed up to 24 months.
  OS was defined as the time from the first dose or random assignment (if any) to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, MD, Principal Investigator — Peking University People's Hospital
Locations (11):
- China (11):
  - Peking University People's Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Chinese PLA General Hospital of Eastern Theater Command, Nanjing
  - Shanghai 6th People's Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou